CLINICAL TRIAL: NCT05414279
Title: Validation of Serum Sodium Levels Through Capillary Blood Collection Via Finger Prick Compared to Standard Venous Blood Sampling
Brief Title: Validation of Capillary Serum Sodium Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-09422
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Nocturia
Keywords: nocturia; Desmopressin; Hyponatremia; Blood chemical analysis
MeSH Terms: conditions — Nocturia; Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capillary and venous sodium (Other): From each patient a capillary and venous blood sample will be taken in order to determine the sodium level
  Interventions: Diagnostic Test: Sodium determination

INTERVENTIONS:
Diagnostic Test: Sodium determination — Through a single finger prick 10 drops of capillary blood will be drawn. The venous blood sample will be taken through a standard venipuncture. Both samples will be send to the lab for indirect sodium determination

SUMMARY:
Prospective interventional study to determine sodium levels in capillary blood via finger prick. The goal is to determine if this technique is suitable and equal to a standard venous blood collection for the analysis of blood sodium levels.The purpose is to compare both sodium levels to determine if they are equal so the technique can be used in a clinical setting for people who need regular blood collections for the determination of sodium, for example after the start of desmopressin use.

DETAILED DESCRIPTION:
Currently, serum sodium levels are determined by standard venous blood sampling. This method is invasive, painful and a relatively large amount of blood is drawn (5ml). Repeated blood draws are necessary in certain patient groups. If sodium values can be determined on a capillary blood sample instead of a classic venous blood sample, the total blood volume will be smaller. In addition, in the future, the aim is to perform capillary blood sampling at home and to send the sample by courier, thus saving the patient a trip to the doctor's office or a nurse at home.

The aim of this prospective interventional study is to validate the sodium values on a capillary blood sample obtained via fingerstick (250µL). To demonstrate that the obtained values are reliable and clinically useful they will be compared one-on-one with the sodium values determined on a standard venous blood sample. Since it is important to validate a broad range of sodium values, a heterogeneous study population is chosen to obtain sufficient variation.

Patients admitted to the Urology department at UZ Gent will be informed verbally and in writing about the content and purpose of the study. If they are interested in participating, they will be asked to sign the consent form. At the moment the already planned venous blood collection, a capillary blood sample will be taken as well via a finger prick. A number of blood drops (250 µL) are collected in a standard Lithium-Heparin tube and will be collected by lab Maenhout for further analysis. The venous blood sample, which is taken as part of the therapy/diagnosis (independent of the study, standard of care) during admission, is analyzed by the clinical lab of UZ Gent.

The sodium values from the capillary blood draw will be compared with the values from the venous blood draw, with each patient acting as their own control. There is no need to have the venous blood samples analyzed by Labo Maenhout, as the clinical lab of UZ Gent uses the same technique for sodium determination (indirect determination) as Labo Maenhout.

The sodium values obtained through capillary and venous blood sampling will be statistically analyzed using a Passing-Bablok regression model.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years or older
* admitted to the urology ward

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Difference in sodium level between capillary and venous blood samples | 1 hour
  the agreement between capillary and venous sodium measurements, measured by the intra-class correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East-Fanders, Belgium

IPD SHARING:
Plan to Share IPD: No